CLINICAL TRIAL: NCT00385957
Title: Comparison of Antiretroviral Activity and Immunological Effect of Two Triple Treatments With and Without Protease Inhibitors in naïve HIV-1-infected Patients With CD4 < 100/mm3
Brief Title: Immunological and Viral Response to Antiretrovirals in HIV Patients With CD4 Cell Count Below 100
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVAN-Z
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2006-10

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: AZT+3TC+IDV+RTV
Drug: AZT+3TC+EFV

SUMMARY:
The study analyzes the virological response in plasma and non-plasma compartments, as well as the degree and kinetics of immune reconstitution in 70 treatment-naive patients with CD4 < 100/mm3, when they receive treatment with two nucleoside analogs (NRTI) plus one protease inhibitor (PI) compared with 2 NRTI plus one non-nucleoside (NNRTI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HIV-1 infection.
* Age 18 years or over.
* No previous antiretroviral therapy.
* CD4 lymphocyte count of < 100 cells/mL.
* Patients who, sufficiently informed, give their written consent to participate in the study and undergo the tests and explorations involved in the study.

Exclusion Criteria:

* Pregnant women, women who are breast feeding, or women who intend to become pregnant during the study period.
* Currently undergoing treatment for an opportunistic infection (parenteral administration).
* Any formal contraindication to treatment with the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70

PRIMARY OUTCOMES:
Proportion of patients with VL below 20 copies/ml in plasma at 12 and 24 months.
Proportion of patients with a CD4 count higher than 200 cells/ml at 12 and 24 months.

SECONDARY OUTCOMES:
Immunophenotypic response at 12 and 24 months (CD4:CD8 quotient,levels of naive
CD4 cells (CD45RA+CD45RO-) and memory cells (CD45RA-CD45RO+)
and levels of CD8 cells (CD28+ y CD38+)
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Gatell, MD, Study Chair — Hospital Clinic of Barcelona
Locations (6):
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - CSU Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Donostia Ospitaleak, Donostia / San Sebastian, Giputzkoa
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Miro JM, Manzardo C, Pich J, Domingo P, Ferrer E, Arribas JR, Ribera E, Arrizabalaga J, Lonca M, Cruceta A, de Lazzari E, Fuster M, Podzamczer D, Plana M, Gatell JM; Advanz Study Group. Immune reconstitution in severely immunosuppressed antiretroviral-naive HIV type 1-infected patients using a nonnucleoside reverse transcriptase inhibitor-based or a boosted protease inhibitor-based antiretroviral regimen: three-year results (The Advanz Trial): a randomized, controlled trial. AIDS Res Hum Retroviruses. 2010 Jul;26(7):747-57. doi: 10.1089/aid.2009.0105. PMID 20624069